CLINICAL TRIAL: NCT00424684
Title: Comparison of the Quantiferon®-TB GOLD (in Tube) Assay With Tuberculin Skin Testing for Detecting Latent Tuberculosis Infection in Patients With Chronic Liver Disease Being Evaluated for or Awaiting Liver Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to obtain contract with sponsor
Sponsor: University of Pittsburgh (Other)
Collaborators: Cellestis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB#0611163
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2015-12

CONDITIONS: Chronic Liver Disease; TB
Keywords: TB; Chronic Liver Disease

INTERVENTIONS:
Procedure: collection of blood sample

SUMMARY:
Tuberculosis (TB) is an important cause of morbidity and mortality in organ transplant recipients. Management of tuberculosis in this setting is challenging due to the complexity of diagnosis and the potential toxicity of anti-TB therapy, especially in liver transplant candidates and recipients. Although the tuberculin skin test (TST) is recommended for screening of latent tuberculosis infection (LTBI) in all candidates for liver transplantation, the performance of the TST in this setting is less than optimal, due to a lack of specificity (false-positive results due to interaction with BCG vaccine and other mycobacterial infections), and a lack of sensitivity in a population that is relatively immunocompromised. Recently, a new test named QuantiFERON-TB Gold (QFT-G) has been approved for the diagnosis of LTBI. QFT-G detects the release of interferon-gamma (IFN-γ) by sensitized white cells after incubation of whole blood with TB antigens. QFT-G is expected to be more specific than TST. However, there are no studies defining the performance of QFT-G in a population of patients on a waiting list for liver transplantation. We plan to estimate the usefulness of the QFT-G test for the diagnosis of LTBI in a cohort of patients with end-stage liver disease. We hypothesize that the QFT-G test will correlate better with the risk of LTBI. This study advances research on the prevention of a serious bacterial infection that can have devastating consequences in the post-transplant setting. The new diagnostic strategy may more accurately determine the presence of LTBI, thereby allowing appropriate therapy.

DETAILED DESCRIPTION:
* Review and record the results of the test/procedures (x-rays, CT-scans, etc.) that are part of the subject's clinical care and the results will become part of the research record. In addition, laboratory results (liver function tests, chemistry, CBC with diff, PT and INR or PTT) will be collected from the medical record.
* Record the list of medications the subject is taking. Collect information on demographics (address, phone number, etc.) including gender, race and ethnicity.
* Review and record past medical and social history

The screening procedures will take a total of about 15-30 minutes and all subjects will be seen in the Liver Transplant Clinic. The investigator and research coordinators will be reviewing the subject's medical record to collect the required information about the subject's medical history. We will ask the subject, if it cannot be found in the medical record, about past TB exposure and treatment, overseas travel, and current resident status (long term care facility, home, hospital, etc.)

If the subject qualifies for the research study the subject will undergo the experimental procedures listed below. These procedures will take place during the visit in the Liver Transplant Clinic.

As part of the liver transplant evaluation subjects will have blood withdrawn for different types of testing. When the blood is obtained we will collect about 3cc of blood for the new TB testing. This collection of the blood sample will occur while the subject is getting their required pre transplant blood work so that they will not need to get stuck twice with a needle. The results of this research testing will not be available to the subject or physicians but will be compared.

The QuantiFERON®-TB Gold IT system uses specialized blood collection tubes, which are used to collect whole blood. Incubation of the blood occurs in the tubes for 16 to 24 hours, after which, plasma is harvested and tested for the presence of IFN-g produced in response to the peptide antigens.

The QFT-G (IT) assay will be performed according to the manufacturer's instructions (Cellestis Ltd.). One mL of whole blood is placed in three separate test tubes, one containing no antigen (nil control), one with TB antigens (ESAT-6, CFP-10 and TB7.7) and one with phytohemaglutinin (mitogen or positive control). The three tubes will be incubated as soon as possible after collection (within 16hrs) and will incubate for 16 to 24 hours at 37°C. Following this incubation period, the tubes will be centrifuged. The plasma will be removed from the tube and placed in a plasma storage container. These containers will then be frozen for future IFN-γ measurement by ELISA. Each institution will perform testing up to this point in the process. Each month, plasma samples will be posted on ice to Edmonton Hospital in Alberta, Canada. The samples will be batched and then undergo the ELISA testing process according to the manufacturer's instructions.

A result of ≥0.35 IU/mL in the TB antigen tube will be considered a positive result. If the level is less than this and the mitogen control is positive (≥ 0.5 IU/mL), a negative result will be recorded. If the level in both the TB antigen and mitogen tube is less than the threshold for positive, then an indeterminate (anergic) result will be recorded. The nil antigen tube adjusts for background IFN-γ levels and is subtracted from the IFN-γ level for the TB antigen and mitogen tube.

Once we have collected the blood sample the subject will have completed the study.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18
* Chronic liver disease on the waiting list or being wait listed for liver transplantation
* Undergoing a PPD test as part of their clinical care

Exclusion Criteria

* Unable to provide informed consent
* Previous history of immediate hypersensitivity to TST
* Previous severe local ulceration with TST
* Suspected active TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01

PRIMARY OUTCOMES:
To assess the concordance between the QFT-G IT assay and the TST in patients with end stage liver disease awaiting liver transplantation and to relate the test results to the patient's risk of latent TB infection.

SECONDARY OUTCOMES:
To assess the factors that are associated with discordance between the TST and the QFT-G test
To assess for laboratory parameters that may influence the QFT-G IT assay, such as lymphocyte count and liver function tests.
To assess the frequency of anergy in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, MD, Principal Investigator — University of Pittsburgh; David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States